CLINICAL TRIAL: NCT05232604
Title: How is Aerobic Exercise Compared to Localized Pain Relief Exercises in Patients With Jaw Pain and Neck Pain? Pilot Study
Brief Title: How is Aerobic Exercise Compared to Localized Pain Relief Exercises in Patients With Jaw Pain and Neck Pain?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hochschule Osnabruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSOS/2020/2/1
Record Dates: First submitted 2021-12-23; First posted 2022-02-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Disorder; Neck Pain
Keywords: Temporomandibular disorder; Neck pain; Exercise therapy; Motor control exercise
MeSH Terms: conditions — Temporomandibular Joint Disorders; Neck Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups (aerobic exercise group and neck motor control exercise group) will receive the protocol at the same time period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assessors (assessing clinician assessed outcomes) and the statistician will be blinded to group allocation. Participants will be unaware of the hypothesis of this study to decrease performance biases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic exercise group (AE) (Experimental): The session training will be divided into a warm-up, main exercise period, and cool-down, with a total duration of 60 minutes (guided by a PT). The training will be performed on a cycle ergometer, three times per week for 12 weeks. The duration of the main AE will be between 30-45 minutes and the intensity will be based on the maximal heart rate (HRmax), heart rate reserve (HRR), and the Borg Rating of Perceived Exertion Scale (Borg Scale), which will be monitored. The intensity of the AE program will be progressively increased according to each patient's response and tolerance but will be standardized as much as possible: 1) first two weeks, low to moderate intensity (60% HRmax or 9-11 on the Borg scale); 2) 2-6 weeks, moderate-intensity (55-70% HRmax or 12-14 on the Borg scale), and 3) last 6 weeks, high intensity interval training (HIT) (75-90% HRmax or 15-17 on the Borg scale; 4 min*4 times HIT followed by 3 min of 70%HRmax in between) will be targeted per literature endorsements.
  Interventions: Other: Aerobic exercise
- Neck motor control exercise group (Active Comparator): The treatment will consist of a 12-week progressive exercise program targeted to the neck flexor and extensor muscles supervised by a physical therapist (PT). This exercise protocol has been successfully tested in subjects with NP. Low load craniocervical exercises (nodding) will be performed at early stages (first 6 weeks) guided by visual feedback from a pressure unit. Higher-load neck exercises will be performed at later stages (last 6 weeks). During the first month, subjects will receive 30-45 min of MCTF three times per week, in the second month twice per week, and in the third month once per week. This duration of treatment is commonly used in clinical settings and has proven to be sufficient to improve muscle function, clinical, and brain outcomes.
  Interventions: Other: Neck motor control exercise

INTERVENTIONS:
Other: Aerobic exercise — 30-45 minutes of aerobic exercise in a cycle ergometer will be applied in three different intensities (low, moderate and high) along 12 weeks of treatment.
  Arms: Aerobic exercise group (AE)
Other: Neck motor control exercise — An specific neck motor control exercise targeted to the neck flexor and extensor muscles supervised by a physical therapist will be applied during 12 weeks of treatment.
  Arms: Neck motor control exercise group

SUMMARY:
Musculoskeletal (MSK) disorders are some of the most burdensome health issues in the world and the leading causes of years living with a disability. Between them, jaw pain and neck have been very prevalent among the general population. Subjects with chronic neck and jaw pain present with persistent pain, allodynia, and hyperalgesia, sometimes extending to regions distant from the neck, head, or face, as well as cognitive and motor dysfunction. In addition, both conditions are commonly related to pain in other anatomical regions, and they also might also exhibit a greater risk for pain-associated somatic symptom burden.

The treatment for patients with neck and jaw could involve different techniques in the rehabilitation area. Between them, therapeutic exercise is a cornerstone of MSK disease rehabilitation. Although mechanisms of action for exercise in subjects with pain are not yet understood, therapeutic exercise is widely applied in a variety of painful MSK conditions, such as low back pain, shoulder pain, knee pain, osteoarthritis, and disorders of the cervical and craniofacial regions such as temporomandibular disorders, headaches, and neck pain. Besides its effects on function and health, therapeutic exercise is known to have some pain-relieving effects and specific motor control exercises targeted to the neck can enhance the neural control of the cervical spine in patients with neck involvement such as patients with jaw and neck pain.

Previous studies have demonstrated that treatment directed to the neck may be beneficial in decreasing pain intensity in the masticatory muscles, increasing pain-free mouth opening, and decreasing pain in the head and neck regions in people with jaw pain. In addition, neck motor control exercises have been successful to manage chronic neck pain and cervicogenic headache. Subjects with neck pain and associated disorders receiving neck motor control exercises had a reduction of pain and improved quality of life. Another option that has been explored to relieve MSK pain is aerobic exercise. Aerobic exercise has been used to stimulate the release of pain-relieving peptides in healthy human beings; however, little is known about the analgesic effect of exercise in people suffering from actual musculoskeletal pain. Previous literature found positive results in favor of aerobic exercise for pain relief. However, none of them included patients with jaw and neck-related disorders. Therefore, the aim of the present pilot randomized controlled trial (RCT) is to test the effectiveness of local craniocervical motor control exercises when compared with aerobic exercise on pain-disability related outcomes such as pain intensity, pain pressure thresholds (PPTs), jaw and neck disabilities and to restore normal muscular performance and fatigability of the cervical muscles in people with jaw and neck pain. Also, an important objective for performing this pilot study is to test the feasibility of these protocols and gather data that will be the basis for applying to external funding.

This study will be a randomized controlled trial, blinded, two-armed parallel group. It will include women between 18-60 years of age; diagnosed with temporomandibular disorders (i.e., jaw pain) classified by the new Diagnostic Criteria for Temporomandibular Disorders (DC/TMD); or diagnosed with idiopathic chronic neck pain associated or not with TMD. Because this is an exploratory (pilot) study it will include at least 21 subjects per treatment group. The primary outcome will be pain intensity evaluated by the Visual Analogue Scale (VAS), and the secondary outcomes will be Neck Disability Index; Jaw Function; Pressure Pain Threshold; Psychological functioning; Global Rating Scale; and Muscular performance and fatigability of the cervical muscles. The patients will be randomized into two groups: local craniocervical motor control exercises and aerobic exercise. The local craniocervical motor control exercises program will be focused on training the deep and superficial flexors and extensors neck muscles. The treatment will consist of a 12-week progressive training program with a total duration of 30-45 min per session. Individuals assigned to the aerobic exercise will receive cycling exercise, with a total duration of 60 minutes. Both groups will be evaluated before the treatment starts (baseline); after two and six weeks from the beginning of treatment (1st and 2nd partial evaluation); at the end of the treatment (final evaluation - 12 weeks); and after three and six months of the end of the treatment (1st and 2nd follow-up).

DETAILED DESCRIPTION:
Musculoskeletal (MSK) disorders are some of the most burdensome health issues in the world and the leading causes of years living with a disability.1 Low back pain, neck pain, and other MSK disorders are within the ten more burdensome conditions in the world. Chronic pain, including chronic MSK pain, is increasing in Europe, and almost one in five Europeans have reported having moderate or severe chronic pain, representing approximately 25-35% of the adult population. Thus, MSK pain is considered a major public health problem due to its high prevalence and considerable burden in terms of medical costs, work disability, and reduced quality of life. The most common MSK pain is located in the back and joints, followed by head and neck pain. Temporomandibular disorders (TMD) or commonly known as jaw pain are one of the chronic musculoskeletal disorders (MSKD) that are in close relationship with neck and head pain and are also considered to be a major public health problem as they are the main source of chronic orofacial pain and the most prevalent category of nondental chronic pain conditions in the orofacial region. These disorders affect the masticatory muscles, the temporomandibular joint, and related structures such as the neck and head.

MSK pain is related to poor individuals´ health status and poor quality of life, affecting the patient's family environment. Specifically, there is abundant evidence that has shown the great impact that neck pain and TMD pain have on the subject's quality of life. They interfere with daily activities, diminishing patient's capacity for work and/or ability to interact with their social environment. Across Europe, around 20% of patients with chronic pain have lost their job or have lost their productivity because of pain; this makes the cost of healthcare very high. In addition, neck pain and TMD have been considered to have a great economic impact due to direct care and have been shown to have similar individual impact and burden as back pain (BP) and severe headache. Therefore, chronic pain, especially musculoskeletal pain has been considered a priority in Europe.

Subjects with chronic neck and jaw pain present with persistent pain, allodynia, and hyperalgesia, sometimes extending to regions distant from the neck, head or face, as well as cognitive and motor dysfunction, demonstrating an abnormal function of the central nervous system similar to other chronic painful conditions. In addition, both conditions are commonly related to pain in other anatomical regions and they also might also exhibit a greater risk for pain-associated somatic symptom burden.

Subjects with neck and jaw pain commonly complain of pain in the neck, face and head region. In a population sample with almost 190000 participants, found that subjects with jaw pain presented generally other pains such as headache, low back pain, and neck pain. Neck pain was one of the most common comorbidities in these subjects. The close relationship between jaw and neck pain and dysfunction has been established by several studies. For example, it was concluded that symptoms of the stomatognathic system overlap in patients with TMD and cervical spine disorder (CSD), and symptoms of the cervical spine overlap in the same group of patients (TMD and CSD). Also, it was found that patients with chronic jaw pain more often suffered from cervical spine pain than those without this disorder. It was found that asymptomatic functional disorders of the cervical spine occurred more frequently in patients with internal derangement of the TMJ than in a control group. The presence of tender points in the cervical and shoulder girdle in patients with the same diagnosis was more common, especially in upper segments of the cervical spine, compared with healthy controls. Also, facial pain was associated with reported pain in the neck area and clinical pain resulting from palpation in the muscles of the neck-occiput area.

Furthermore, the literature has highlighted that people with jaw and neck pain have neck muscle impairments relative to healthy people, specifically abnormalities in endurance and performance of the cervical flexor and extensor muscles. People with jaw and neck pain also demonstrate poor performance in the Craniocervical Flexion Test, with the increased electromyographic activity of the superficial cervical flexor muscles. These results implicate the altered endurance capacity of the flexor and extensor cervical muscles that lead to neck-shoulder disturbances observed in people with jaw and neck pain. These physical impairments seem to be a common factor of subjects with neck pain involvement such as cervicogenic headache, and whiplash-associated disorders.

Therapeutic exercise is a cornerstone of MSK disease rehabilitation. Although mechanisms of action for exercise in subjects with pain are not yet understood, therapeutic exercise is widely applied in a variety of painful MSK conditions, such as low back pain, shoulder pain, knee pain, osteoarthritis and disorders of the cervical and craniofacial regions such as temporomandibular disorders, headaches, and neck pain. Besides its effects on function and health, therapeutic exercise is known to have some pain relieving effects and specific motor control exercises targeted to the neck can enhance the neural control of the cervical spine in patients with neck involvement such as patients with jaw and neck pain.

From our previous studies on neck muscle impairment in people with jaw pain and our recent update of a systematic review on therapeutic exercise to manage jaw pain, it was concluded that neck motor control exercise is a promising option to treat people with these disorders. Studies showed that treatment directed to the neck may be beneficial in decreasing pain intensity in the masticatory muscles, increasing pain-free mouth opening and improve pain in the head and neck regions in people with jaw pain. In addition, neck motor control exercises have been successful to manage chronic neck pain and cervicogenic headache. Subjects with neck pain and associated disorders receiving neck motor control exercises had a reduction of pain and improved quality of life.

Another option that has been explored to relieve MSK pain is aerobic exercise. Aerobic exercise has been used to stimulate the release of pain-relieving peptides in healthy human beings; however, little is known about the analgesic effect of exercise in people suffering from actual musculoskeletal pain. Several systematic reviews looking at different modalities of aerobic exercise for managing MSK pain have been found. These reviews looked at low back pain, knee pain, chronic MSK pain, migraine among others. From all of the studies looking at different MSK conditions, 19 studies compared aerobic exercise to a control group. Among them, five studies found a positive medium and large effect sizes in favor of aerobic exercise for pain relief. However, none of these reviews and their included studies looked at the effectiveness of aerobic exercise for jaw and neck related disorders. Thus, the evidence is still limited. Therefore, these results warranty an RCT with the aim of answering the following questions:

Q1) What is the effectiveness of neck motor control training using visual feedback (MCTF) and aerobic exercise on pain-disability related outcomes such as pain intensity, pain pressure thresholds (PPTs), and jaw and neck disabilities in people with jaw and neck pain? Hypothesis: People with jaw and neck pain receiving neck MCTF will have decreased pain intensity, increased pain pressure threshold, and decreased disability in the neck and jaw after 12 weeks of treatment and 3 and 6 months after treatment ends (between group comparison) when compared with subjects receiving aerobic exercise.

Q2) What is the effectiveness of neck MCTF and aerobic exercise in patients with jaw and neck pain to restore normal muscular performance and fatigability of the cervical muscles? Hypothesis: People with jaw and neck MSK pain receiving MCTF will have positive changes in their jaw and cervical muscular performance and fatigability of the superficial cervical flexor and extensor muscles after 12 weeks of treatment and 4 months after treatment ends (between group comparison) when compared with subjects receiving aerobic exercise.

The aim of the present pilot randomized controlled trial (RCT) is to test the effectiveness of local craniocervical motor control exercises when compared with aerobic exercise on pain-disability related outcomes such as pain intensity, pain pressure thresholds (PPTs), jaw and neck disabilities and to restore normal muscular performance and fatigability of the cervical muscles in people with jaw and neck pain. Also, an important objective for preforming this pilot study is to test the feasibility of these protocols and gather data which will be the basis for applying to external funding.

This study will be a RCT, blinded, two-armed parallel group. Sample size. A convenience sample of subjects with jaw and neck pain who attend any physiotherapy or health related clinic in the city of Osnabrück or surroundings will be recruited for this project. No previous studies comparing motor control exercises and aerobic exercises were found; and thus, there is no explicit effect size to base our calculation on. However, it is anticipated that motor control exercises would be better than aerobic exercises and the effect size would be moderate (ES=0.6) on current pain intensity. It would be run a pilot study which will help generate the estimates for these outcomes for future trials. Although sample size calculation for pilot studies is not crucial, the literature has suggested that pilot sample sizes per treatment arm be at least 15 patients per group if the effect size is medium (0.4-0.7). The literature reports dropout rates of 20%. Therefore, in an exploratory fashion, it will be targeting at least 21 subjects per each treatment group (42 subjects in total due to the possibility of a 20% of dropouts).

Procedure. An experienced assessor will determine subjects' eligibility. Demographic data including age, weight, and height will be also collected. All questionnaires are translated to the German language. In addition, the primary outcome will be pain intensity evaluated by the Visual Analogue Scale (VAS), and the secondary outcomes will be Neck Disability Index; Jaw Function; Pressure Pain Threshold; Psychological functioning; Global Rating Scale; and Muscular performance and fatigability of the cervical muscles. The patients will be randomized into two groups: local craniocervical motor control exercises (group 1) and aerobic exercise (group 2).

Randomization. A randomization sequence stratified by age group (18-30, young adult; 31-45, adult; 46-60, older adult) and condition (jaw pain and neck pain), will be computer-generated by a researcher not involved in the study. The allocation concealment will be done by an assistant, who will distribute the results of the sequence into an electronic platform (Redcap) to ensure the concealment. Patients (unaware of the hypothesis of this study), assessors (measuring the outcomes for this study), and the statistician will be blinded to group allocation following established guidelines.

Treatments. The local craniocervical motor control exercises program will be focused on training the deep and superficial flexors and extensors neck muscles. The treatment will consist of a 12-week progressive training program with a total duration of 30-45 min per session. While Individuals assigned to the aerobic exercise will receive cycling exercise, with a total duration of 60 minutes for 12 weeks.

Timeline. Both groups will be evaluated before the treatment starts (baseline); after two and six weeks from the beginning of treatment (1st and 2nd partial evaluation); at the end of the treatment (final evaluation - after 12 weeks of the beginning); and after three and six months of the end of the treatment (1st and 2nd follow-up).

Compliance and contamination. The compliance and contamination will be controlled through reminders and diaries via RED-Cap. It would be also offer flexible session schedules to fit participant needs. For patients in the motor exercise group, it will be encouraged that participants to follow the protocol at home and require them to record compliance with exercises in a patient diary where they have to register whether they perform the exercises and the amount of them daily. These records will be considered in analyzing the results of the trial by using the compliance as a covariate and by using per-protocol analysis. Participants will be treated individually in a clinic and will be not involved with other participants. In addition, participants will be asked to refrain from other treatments such as physical therapy, new splint therapy, chiropractor during the study to avoid co-interventions. Pain medications already used by the study participants will be allowed, and changes in medications will be monitored by the therapist each visit. Any changes to the trial protocol will be registered by the researchers in REDCap and will be considered in analyses.

Statistical Analysis. Following CONSORT guidelines, the analysis will follow the intention to treat principle. Data will be described for each intervention group (e.g., means, standard deviations). Change scores (all evaluation time minus baseline) will be summarized for each outcome. Separate 2-sample, 2-sided t-tests will assess differences in intervention groups on mean change scores at these evaluation periods for VAS, PPT, TMDs and neck disabilities, and neck performance and fatigability. These analyses may also be repeated using multiple imputation methods in the event of substantive dropout. Additionally, analyses will include separate mixed effects multiple linear regression models for each outcome to assess the effect of intervention over time and adjust by other variables that may not have been balanced across groups by randomization. Model estimates and associated 95% confidence interval (CIs) will be reported and residual diagnostics will assess model fit. Effects sizes (ES) and minimal important difference (MID) of the outcomes (using the GRS as an anchor measure) will be used to determine the clinical significance of the results. R software will be used for statistical analysis by a data analyst, blinded to intervention group.

Positive and negative consequences for the test subjects. Exercises, either targeted to the neck or aerobic exercises could be a simple and conservative way to improve pain and disability for patients with jaw and neck pain. Subjects participating in this study might improve their clinical symptoms and improve their quality of life. It is expected that the results of this study could help clinicians, rehabilitation groups, and scientists to treat patients with jaw and neck pain in a more effective way. There are no known negative consequences for test subjects with these exercise protocols. However, if some negative consequences arise the appropriate steps will be taken. Payment to participants will not be provided due to the lack of funding for this study.

Planned measures for crisis intervention for the possible injuries/damage. Injuries related to these protocols are not known, so it is not expected that this should happen. However, it is possible that someone feels muscle soreness at the evaluation time points or at the beginning of the training sessions, especially for sedentary participants. This soreness will most likely disappear in a few days and will not cause major damage to the patient. However, if the soreness persists the patients will be instructed to perform stretches, use cold or heat and take a rest period. If nevertheless, the symptoms persist, it will be suggested that the patient consults a physician.

Measures to ensure data protection and data security (Storage of the data). All data will be kept private, under protection in a safe area, and just could be open when required by law. All data will be kept at least five years after the end of the study. The name or any other identifying data from the participant will not be attached to the data. These identification data will never be used in any publication or presentation. Before the data analyses, all ethical principles will be reviewed to ensure that the data are used ethically. The researcher will explain all procedures to the participants to ensure that they are aware of the researchers 'responsibilities regarding privacy and confidentiality. To guarantee the anonymization of data, all participants will receive an identification code, then their personal data (especially, their names) will be reserved and be secured.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-60 years of age
* Be diagnosed with idiopathic chronic neck pain as described the IASP and/or presence of temporomandibular disorders identified by DC/TMD screening
* Have pain in the neck or jaw area for at least 3 months (chronic pain)
* Have pain not attributable to recent acute trauma, previous infection, or to an active inflammatory cause in the last month
* Have a moderate or severe baseline pain score of 30mm or greater using a 100mm VAS

Exclusion Criteria:

* Present red flags for serious pathologies related to neck pain or jaw pain
* Report comorbidity functional chronic pain disorders (e.g., fibromyalgia)
* Have been diagnosed with psychiatric disorders (e.g., depression, schizophrenia)
* Have received therapy within 3 months prior to entry into the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Analog Scale (mean change at 12 weeks) | Main Outcome is pain change at 12 weeks. Other time points will also be collected (baseline, 2, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  A change in pain intensity (measured with the VAS) from baseline to end of treatment (12 weeks) for both groups. The pain evaluated will be the pain related to the patient's main complaint, i.e. jaw pain or neck pain. The VAS is a 100 mm linear scale, labeled with the two extreme boundaries of pain sensation: "no pain" at one end (0 mm) and "worst pain imaginable" at the other end (100 mm). The VAS has demonstrated validity and reliability to measure the intensity of pain and it is heavily used in people with neck pain as well as jaw pain research. The VAS varies from 0 to 100 mm, and the higher values means worse results.

SECONDARY OUTCOMES:
Neck Disability Index | baseline, 2, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  It is a 10-item questionnaire that measures how much neck pain affects activities of daily living. The Neck Disability Index (NDI) is a validated, reliable and responsive tool. The scores varies from 0 to 50 points, and the higher values means a worse result.
Jaw function scale | baseline, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  It will be measured using a self-reported questionnaire called Jaw functional limitation scale form the DC/TMD instruments. This tool has been shown to be valid and has excellent psychometric properties. The total score will be used for statistical purposes. The scores varies from 0 to 50 points, and the higher values means a worse result. The scores varies from 0 to1 points, and the higher values means a worse result.

OTHER OUTCOMES:
Mouth range of motion | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  All mouth range of motion will be measured: maximal mouth opening (MMO), lateral excursion to the right and left, and protrusion with a digital caliper tool. There is no specific range of values to be obtained, but all measures will be measure in millimetres (mm), and higher values means a better result.
Upper and global Neck range of motion | baseline, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  Upper neck range of motion (ROM) will be measured by performing the Flexion Rotation test to the right and left. All global neck range of motion will be measured: flexion, extension, lateral-flexion and rotation. All measures will be done with a Neck care device. There is no specific range of values to be obtained, but all measures will be measure in degrees, and higher values means a better result.
Pressure pain threshold | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  Pressure pain sensitivity will be evaluated via pressure pain threshold (PPT), or the minimum pressure that induces pain or discomfort. This will be done in the masticatory muscles and neck muscles using a calibrated mechanical algometer following the protocol described in Silveira et al. PPT measurements have been shown to have good or excellent inter-rater and intra-rater reliability (0.74 to 0.99). There is no specific range of values to be obtained, but all measures will be measure in Newtons (N), and higher values means a better result.
Heart Rate | baseline, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The maximal heart rate (HRmax) will be calculated through the modified Bruce´s Protocol or by the ramp protocol for cycle ergometer. The modified Bruce´s Protocol is a treadmill test where the speed and the slope of the treadmill are increased systematically every three minutes. The first stage starts with 1.7 mph or 2.7 km/h without inclination of the treadmill for three minutes. Then, the second stage is done with a speed of 2.7 km/h with a slope of 5%. The test ends when the patient reports fatigue. Usually, the ramp protocol for cycle ergometer uses increments of the intensity of 5 to 50 w/minute to measure the HRmax, depending on the functional capacity of the participant. These increments could be determined for women by the formula proposed by Wasserman et al: [(height in cm - age) x 20] - [150 + (6 x weight in kg)]/ 100. There is no specific range of values to be obtained with this test.
Craniocervical flexion test (CCFT) | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  To test the performance of the deep cervical muscles. To perform the test, the volunteer will lay in supine with the neck in a neutral position and with biofeedback placed behind the neck in the occipital area inflated to a baseline of 20 mmHg the patient will be instructed to perform a movement gently and slowly as a "yes" head-nodding action. The test presents 5 progressive levels with a 2mmHg for the biofeedback equipment, based on that the pressure will range from 20mmHg to 30mmHg. The patient should perform as much they can of 10 repetitions with 10 seconds of duration in each. The scores varies from 20 to 30 mmHg, and the higher values means a better result.
Neck extensor endurance test | baseline, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The volunteer is placed in prone lying with the arms at their side and the head over of the end of the plinth. The test person is additionally restrained by three Velcro straps. The first fixes the chest and cervicothoracic junction on the plinth and the second the pelvis. The participant is instructed to do an extension of the neck against a dynamometer maintaining 25% of the maximal voluntary contraction (MVC). If the test person can no longer maintain the specified performance level of 25%, i.e. deviates conspicuously from the reference lines and does not manage to maintain the performance again even after correction, the test is terminated. Another termination criterion is fulfilled if the test person decides independently to end the test because of pain or discomfort. There is no specific range of values to be obtained, but the time of the test is counted in seconds, and higher values means a better result.
Neck flexor endurance test | baseline, 6 weeks after the beginning of treatment, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The volunteer lays in a supine position and with the head positioned, by the therapist, in a slight upper neck flexion on the therapist hand below the occiput. Then it is requested to the volunteer to flex the lower neck and lift the head off the therapist's hand while keeping the upper neck flexion and maintaining a 25% of the maximal voluntary contraction measured with a dynamometer. The test is finalized when the volunteer can no longer maintain the specified performance level of 25%, i.e. deviates conspicuously from the reference lines and does not manage to maintain the performance again even after correction, the test is terminated. Another termination criterion is fulfilled if the test person decides independently to end the test because of pain or discomfort. There is no specific range of values to be obtained, but the time of the test is counted in seconds, and higher values means a better result.
Psychological functioning (distress) | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The distress will be measured by the patient health questionnaire-15 (PHQ-15) recommended by the DC/TMD such as the for distress. This questionnaires are all validated to be used in patients with TMD. The scores varies from 0 to 30 points, and the higher values means a worse result.
Psychological functioning (depression) | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The depression symptoms will be measured by the patient health questionnaire-9 (PHQ-9) recommended by the DC/TMD. These questionnaires are all validated to be used in patients with TMD. The scores varies from 1 to 27 points, and the higher values means a worse result.
Kinesiophobia (Tampa Scale) | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The kinesiophobia will be measure by the Tampa Scale of Kinesiophobia. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia. So, higher values means a worse result.
Kinesiophobia (Neck Pix) | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The kinesiophobia will be measure by the NeckPix which was designed to measure the beliefs of subjects with chronic non-specific NP concerning pain-related fears of a specific set of ADL's in such a way that the scale score would generalise to a measure of activity-related kinesiophobia. In completing the Neck-Pix©, subjects are asked to rate each picture from 0 (no fear) to 10 (greatest fear) according to the question: How much do you fear doing this activity would hurt your neck?, and the scale total score (0-100) is expected to generalise to a measure of activity-related kinesiophobia.
  So, higher values means a worse result.
Level of chronic pain | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The level of chronic pain will be measure with the Graded Chronic Pain Scale. The scores varies from 1 to 3 scale score, and the higher values means a worse result.
Quality of pain | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  To assess the severity of pain and its impact on functioning the Brief Pain Inventory will be used. The scores varies from : 1 - 4 = Mild Pain; 5 - 6 = Moderate Pain and, 7 - 10 = Severe Pain. The higher values means a worse result.
Central sensitization | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  Central sensitization Inventory (CSI) is an instrument to assess somatic and emotional complaints associated with central sensitization syndrome. The questionnaire is composed of part A with 25 questions related to health symptoms and part B which collects information about to previously diagnoses. This tool can quantify the severity of the symptoms and demonstrated to be statistically valid and clinically useful. The higher values means a worse result.
Fear avoidance | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  Fear avoidance is a questionnaire composed of two subscales based on the patient's belief of how the pain affects physical activity and work. This tool is used in clinical practice in order to identify patients with a risk of prolonging disability because of high fear avoidance beliefs. This questionnaire was translated for the German language and present good reliability, and validity. The 7-item work scale has a point score that ranges from 0-42 points. The higher values means a worse result.
Quality of life: General | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The quality of life will be measured by three questionnaires. The 36-Item Short Form Healthy Survey (SF-36) which is a valid self-response questionnaire widely used to measure the health-related quality of life (HRQoL). The questionnaire presents two independent constructs physical and mental health and assesses eight health concepts (physical functioning, role limitations because of physical health problems, bodily pain, social functioning, general mental health, role limitations because of emotional problems, vitality and general health perceptions) in 36 questions. The higher values means a better result.
Quality of life: Oral | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The quality of life will be measured by the Limitation of daily function questionnaire which it was designed to provide information about the extent to which the jaw affects the ability to manage daily life in patients with jaw pain. The higher values means a better result.
Quality of life: Oral | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  The quality of life will be measured by the Oral Health Impact Profile (OHIP-14) which is a questionnaire specific to test the quality of life of patients with orofacial pain. The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse and lower scores indicate better oral health quality of life.
Oral Behaviors Checklist | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  Oral Behaviours Checklist is a self-report scale for identifying and quantifying the frequency of jaw overuse behaviours. The higher values means a worse result.
EQ-5D questionnaire | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  EQ-5D is a self-reported instrument developed to be used in health care evaluation based on five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be answered on a five points scale. A second part is a thermometer rating with a VAS scale from 0 (worst health the patient can imagine) to 100 (best health the patient can imagine) for the individual rating your own healthy. This tool has been validated for the German language. The higher values means a worse result.
Credibility and Expectancy Questionnaire (CEQ) | After 1 day of treatment
  Credibility and Expectancy Questionnaire (CEQ) is a questionnaire that presents two sections related to what the patient thought and fell about the treatment. This questionnaire shows high internal consistency and good reliability. There is no specific values to be obtained.
Level of physical activity | baseline, final evaluation (12 weeks after the beginning of treatment), three and six months after the end of treatment
  International Physical Activity Questionnaire long version (IPAQ) is a self-reported questionnaire with good validity and reliability. The tool is composed of 31 questions that questions evaluate four domains of physical activity: occupation, transport, household and leisure time. The higher values means a better result.

CONTACTS AND LOCATIONS:
Locations (1):
- Hochschule Osnabrück - University of Applied Sciences, Osnabrück, Lower Saxony, Germany